CLINICAL TRIAL: NCT06336174
Title: Cognitive Decline and Underlying Mechanisms in Symptomatic Intracranial Atherosclerotic Stenosis Patients: A Multicenter Cohort Study
Brief Title: Cognitive Decline and Underlying Mechanisms in Symptomatic Intracranial Artery Stenosis Patients: A Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head of Neurology, Principal Investigator，Clinical Professor, Anhui Medical University
Other Study IDs: Anhui-SIA-cohort
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Atherosclerosis; Cognitive Impairment; Cerebrovascular Event
Keywords: Symptomatic Intracranial Atherosclerosis Stenosis; Cognitive Impairment; Cerebravascular Event
MeSH Terms: conditions — Intracranial Arteriosclerosis; Cognitive Dysfunction | interventions — Aspirin; Clopidogrel; Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and anticoagulant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery Group: Symptomatic intracranial stenosis patients who receive endovascular therapy combined with standard medical treatment
  Interventions: Procedure: Endovascular therapy,Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin
- Medical group: Symptomatic intracranial stenosis patients who receive standard medical treatment without endovascular therapy
  Interventions: Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin

INTERVENTIONS:
Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin — All patients received standard medical management, including dual antiplatelet therapy (aspirin and clopidogrel) for three months with aspirin or clopidogrel monotherapy thereafter and high-dose statin, and treatment of hypertension to guideline targets.
  Groups: Medical group
Procedure: Endovascular therapy,Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin — All patients underwent endovascular therapy and received standard medical management after surgery, including dual antiplatelet therapy (aspirin and clopidogrel) for three months with aspirin or clopidogrel monotherapy thereafter and high-dose statin, and treatment of hypertension to guideline targets.
  Groups: Surgery Group

SUMMARY:
The purpose of this study is to explore the mechanism of cognitive impairment in patients with symptomatic intracranial atherosclerotic stenosis (ICAS), and further plans to explore the impact of different treatment options on cognitive function in symptomatic ICAS patients.

DETAILED DESCRIPTION:
All participants underwent a medical evaluation that included routine laboratory studies before and after 3-month and 1-year follow-up. Upon meeting the inclusion criteria and providing informed consent, each participant will complete a battery measure of neuropsychological tests, blood sample collection, and magnetic resonance imaging scan after enrollment and after 3-month and 1-year follow-up.

About 100 participants were included in this study. A series of neuropsychological tests were obtained by a trained investigator to assess. The tests include the evaluation of global cognitive function and multiple individual cognitive domains. The various tasks and questionnaires to measure cognition function including Montreal Cognitive Assessment (MoCA), Mini Mental State Examination (MMSE), Chinese Auditory Verbal Learning Test (CAVLT), Digital Span Test (DST), , Stroop color test (Stroop test), Color trail test (CTT), Clock Drawing Test (CDT), Verbal Fluency Test (VFT), etc., at the same time, the investigators also pay attention to the evaluation of participants' emotions by Hamilton Anxiety Scale (HAMA), Hamilton Depression Scale (HAMD). Furthermore, the memory and the occurrence of cerebrovascular events as the primary outcome measure, this study focused on the multidimensional cognitive function and cerebrovascular events of patients with symptomatic ICAS. Blood sample will be collected for biological multiomics research. The patients will receive a magnetic resonance imaging scan in multi-modalities.

After 3-month and 1-year follow-up, the participants will be interviewed to obtain the same assessments, blood sample and magnetic resonance imaging scan in multi-modalities as before.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Severe stenosis (≥70%-99%) of atherosclerotic internal carotid artery (C6 segment, C7 segment) or middle cerebral artery (M1 segment) confirmed by digital subtraction angiography (DSA) or at least two of the following non-invasive examinations: magnetic resonance angiography (MRA), computed tomography angiography (CTA), or transcranial Doppler (TCD)
* Transient ischemic attack (TIA) or minor stroke (National Institute of Health Stroke Scale [NIHSS] score ≤ 4 points)
* Right-handed and able to cooperate in neuropsychological tests
* At least 14 days post-onset of cerebral infarction or TIA
* Signed informed consent

Exclusion Criteria:

* Other diseases that affect cognitive function, such as cerebral hemorrhage, •Parkinson's disease, neurosyphilis, dementia, tumors, etc.
* Right upper limb hemiplegia, aphasia, visual field defects, or visual impairments
* More than 50% stenosis of the extracranial internal carotid artery, the vertebral artery, or the basilar artery
* Vasculitis, moyamoya disease, and cardiogenic stroke
* Previous history of head and neck stent implantation, carotid endarterectomy, aneurysm embolization, or other intracranial surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial stenosis which was defined as stenosis of 70% or more in Intracranial segment of internal carotid artery and middle cerebral artery (MCA) with transient ischemic attack or minor stroke(NIHSS≤4 points).The degree of stenosis was measured by transcranial doppler, computed magnetic resonance angiography (MRA),tomography angiography (CTA) and digital subtraction angiography (DSA).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in Memory | baseline, 3-month and 1-year follow-up
  The changes in Memory function will constitute one of the main indicators of research results, which will be used to evaluate the follow-up results of the standard treatment regimen. The investigators will use the Chinese Auditory Verbal Learning Test (CAVLT) to evaluate the immediate, delayed and recognition memory of patients with symptomatic ICAS to evaluate the immediate, delayed and recognition memory of patients with ICAS.
Occurrence of ischemic cerebrovascular events | baseline, 3-month and 1-year follow-up
  The changes in occurrence of ischemic cerebrovascular events constitute another major indicator of research result. The new responsible cerebrovascular events during the follow-up period are also the clinical information the investigators pay attention to, including transient ischemic attack (TIA) and stroke.

SECONDARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | baseline, 3-month and 1-year follow-up
  The changes in MoCA will constitute the secondary research outcome. MoCA was based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. The investigators adopted a localized version (Mandarin-8.1 version) in line with the Chinese cultural background. It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better.
MMSE (Mini Mental State Examination) | baseline, 3-month and 1-year follow-up
  The changes in MMSE will also constitute the secondary research outcome. The full name of MMSE is mini-mental state examination, and the scale consists of 30 subjects, include the following seven aspects: time orientation, place orientation, immediate memory, attention and calculation, delay memory, language, visual space. One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answer he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, the investigators suspect that scores would decrease after follow-up.
DST (Digital Span Test; Forward and Backward) | baseline, 3-month and 1-year follow-up
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward (0-14) and backward (0-13). In the forward test, the subjects were asked to retell the the digits immediately after hearing it until they could not be repeated correctly. In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better. In this study, the investigators suspect that scores would decrease after follow-up.
The Stroop Color Test | baseline, 3-month and 1-year follow-up
  The changes in The Stroop color test will constitute the secondary research outcome measure. The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects
CTT (Color Trail Test) | baseline, 3-month and 1-year follow-up
  The changes in CTT will constitute the secondary research outcome. The Color Trail Test (CTT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.In this study, the investigators suspect that scores would decrease after follow-up.
CDT (Clock drawing test) | baseline, 3-month and 1-year follow-up
  The clock drawing test is currently widely used in the evaluation of cognitive impairment, requiring a free hand drawing of a clock within 10 minutes with the pointer pointing towards 11:10, which can be well used to evaluate the visual spatial ability of participants. The commonly used scoring methods include the 3-point method, the 4-point method, and the 10-point method.
VFT (Verbal Fluency Test) | baseline, 3-month and 1-year follow-up
  The changes in The Verbal Fluency Test (VFT) will constitute the secondary research outcome measure. The VFT can be used to evaluate the frontal lobe fluency of patients, mainly including semantic verbal fluency and phonemic verbal fluency.
HAMD (Hamilton Depression Scale) | baseline, 3-month and 1-year follow-up
  The changes in HAMD will constitute the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms.
HAMA (Hamilton Anxiety Scale) | baseline, 3-month and 1-year follow-up
  The changes in HAMA will constitute the secondary research outcome. Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety.
MRI measure- resting state MRI images | baseline, 3-month and 1-year follow-up
  The resting state magnetic resonance data were collected to compare the neuroimaging differences between the patients and healthy control groups.
MRI measures-structural phase MRI images | baseline, 3-month and 1-year follow-up
  The structural phase magnetic resonance data were collected to compare the neuroimaging differences between the patients and healthy control groups.
MRI measures-3D pCASL images | baseline, 3-month and 1-year follow-up
  The three-dimensional pseudo continuous Arterial Spin Labeling (3D pCASL) data were collected to compare the differences in cerebral perfusion between the patients and healthy control groups.
Ultrasound measures-MCA-PI (middle cerebral artery-pulsatility index) | baseline, 3-month and 1-year follow-up
  Pulsatility index (PI) in the middle cerebral artery (MCA) is considered a measure of peripheral vascular resistance. The investigators want to explore the peripheral vascular resistance by MCA-PI.
Ultrasound measures-IMT (intima-media thickness) | baseline, 3-month and 1-year follow-up
  The carotid intima-media thickness (IMT) is a widely used surrogate marker for atherosclerosis worldwide. The investigators want to explore the risk of recurrence of cerebrovascular events by IMT.
Blood Metabolomics measures-CRP (C-reactive protiein) | baseline, 3-month and 1-year follow-up
  CRP is a plasma protein synthesized by the liver and is often used as a nonspecific biomarker of inflammation. Elevated CRP levels are associated with increased risk of cerebrovascular disease and dementia. The investigators intend to use CRP to explore the relationship between inflammatory response and cognitive impairment.
Blood Metabolomics measures-oxLDL(Oxidized low-density lipoprotein) | baseline, 3-month and 1-year follow-up
  Oxidized low-density lipoprotein (oxLDL) is a biomarker that is a key factor for the occurrence and development of atherosclerosis and the formation of unstable plaque. Atherosclerosis has been associated with the onset, severity and progression of cognitive dysfunction. The investigators intend to further explore the relationship between LDL level and cognitive impairment.
Blood Metabolomics measures-miRNA/microRNA | baseline, 3-month and 1-year follow-up
  microRNA (miRNA) is a type of non-coding single-stranded small RNA that plays a role in biological functions by regulating post-transcriptional gene expression. miRNA is involved in the regulation of synaptic plasticity and is related to learning and memory. The investigators intend to reserve serum samples for the study of miRNA and cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China